CLINICAL TRIAL: NCT01281345
Title: A Multicenter Observational Study of Candidemia Among ICU Patients in India
Brief Title: SIHAM Candidemia Network:An Observational Study
Status: Completed | Type: Observational
Sponsor: Society of Indian Human & Animal Mycologist (Other)
Responsible Party: Principal Investigator, Prof. Arunaloke Chakrabarti, Professor, Society of Indian Human & Animal Mycologist
Other Study IDs: SIHAM_02
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2011-01

CONDITIONS: Candidemia
Keywords: icu; candida; epidemiology; blood stream infection; candidemia
MeSH Terms: conditions — Candidemia; Torulopsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Candida isolates
Oversight: Data Monitoring Committee: No

SUMMARY:
Title: A multicenter observational study of candidemia cases among ICU patients in India

Objective: Primary objective:

Determine epidemiological and also clinical parameters of candidemia cases among ICU patients in India.

Exploratory Objectives:

1. Determine the prevalence of candidemia among ICU patients.
2. Determine the prevalence of candidemia due to C. albicans and each species of non-albicans Candida species.
3. Determine the demographics and risk factors for candidemia patients and comparison of relevant variables between the cases with C. albicans and non-albicans Candida species isolation.
4. Describe physician practice in the management of candidemia cases - clinical and outcome.
5. Determine the in-vitro antifungal susceptibilities of Candida isolates.

Study description and purpose:

Short description: Observational multicentre study in ICU patients. Study purpose: Epidemiological determinants of candidemia, management and outcome evaluation.

How the study would help? It would help to evaluate outcomes of current management strategies and to develop future better management strategies of candidemia cases.

Critical issues & risk: Site & center selection would be important No risk for patients included in the study as it is only observational study

Study design:

Site selection: A questionnaire will be circulated (annexure I) to all major tertiary care centers of India. The centers will be selected on the competence of candidemia diagnosis and availability ICU facilities. Expected number of centers ~ 20.

Study period: October 1, 2010 - March 31, 2012 No of patients/sites: Consecutive all patients with candidemia detected during ICU stay over the study period will be included in the study in each site.

Patient selection: Inclusion criteria:

1. Admitted in ICU for > 48 hours (to coincide definitions of nosocomial or ICU-acquired)
2. All age group patients will be included (pediatric & adult)
3. Diagnosed as proven candidemia (isolation of Candida species from blood culture on ≥ 1 occasion during ICU stay)
4. Blood culture positive for Candida spp. , if sample has been drawn within 48 hrs after discharge from the ICU.

Exclusion criteria:

1. Patient already diagnosed of candidemia before admission in ICU Variables|: types of ICU, demographic data of patients, underlying illness, risk factors, severity scores, diagnostic methods, treatment characteristics (Annexure II) and treatment outcomes (Annexure III)

Diagnosis of candidemia: Isolation of Candida species from blood culture (arterial/venous) by any method (conventional/ lysis-centrifugation/ automated system/ any other method). No intervention in diagnostic processes at any center. Centers not performing diagnosis of candidemia will be excluded from the study

Data recording: both manual and online. The form of Annexure II will be filled up within 5 days of diagnosis of candidemia; Annexure III will be filled up within 7 days of discharge from hospital or 30 days after starting the antifungal therapy or death of the patient (which over period is early).

Data analysis: appropriate statistical method will be employed for analysis of data.

DETAILED DESCRIPTION:
1. Objectives :

   1.1. Primary objective: Determine the epidemiological parameters of candidemia cases among ICU patients in India 1.2. Exploratory objectives
   1. Determine the prevalence of candidemia among ICU patients.
   2. Determine the prevalence of candidemia due to C. albicans and each species of non-albicans Candida species.
   3. Determine the demographics and risk factors for candidemia patients, and comparison of relevant variables between the cases with C. albicans and non-albicans Candida species isolation.
   4. Describe the management of candidemia cases and outcome.
   5. Determine the in-vitro antifungal susceptibility testing of Candida isolates.
2. Study description and purpose:

   2.1 Observational multicentre study of ICUs in India. Institute having ICUs and facility for diagnosis of candidemia will be chosen.

   2.2 Purpose: Determination of epidemiological parameter of candidemia, description of current management and outcome of patients with candidemia. This would help in formulation of a guideline for management of patients with candidemia especially when the patients are critically ill and admitted in ICUs.

   2.3 Critical issues & risk: There is no risk for patient as it only observational study and no intervention is intended. The site selection would be important to get useful data.
3. Study design:

   3.1 Site selection: The major tertiary care centers will be evaluated on the basis of responses to a set of questionnaire (Annexure I). Only centers having ICU facilities and competence to diagnose candidemia will be selected. Expected number centers will be ~20.

   3.2 Study period: October 1, 2010 - March 31, 2012

   3.3 No of patients: Consecutive patients with candidemia diagnosed in ICUs > 48 h after admission during the study period will be included in each site. Expected number of patients with candidemia would be ~2000
4. Patient selection:

   4.1 Inclusion criteria:
   1. Admitted in ICUs for > 48 hours
   2. All age group patients will be included (both adult & children)
   3. Diagnosed as proven candidemia with isolation of Candida species ≥1 occasion from blood during ICU stay.
   4. Blood culture positive for Candida spp. , if sample has been drawn within 48 hrs after discharge from the ICU.

   4.2 Exclusion criteria: a) Patient already diagnosed for candidemia before admission in ICUs or in ICU for ≤48h .
5. Patient management:

   During the study period, all process of patient management including diagnosis and treatment will be determined by treating physician. There will be no intervention in patient management as a part of study related activities.
6. Conduct of the study 6.1 Investigators of the study - The ICU specialist in charge and microbiologist/mycologist of each center will be the site investigators of the study. Prof. Arunaloke Chakrabarti of PGIMER, Chandigarh will be coordinator of the study. A/Prof. Sharon Chen, Medical Mycologist, Infectious Diseases and Microbiology, Westmead Hospital, Australia will be the advisor of the study.

6.2 Patient enrollment - The investigator should ensure that only the patients with candidemia development in the ICU (see inclusion criteria) are included. Consecutively all patients meeting the eligibility criteria will be consecutively enrolled. The patients will be enrolled prospectively as soon as the diagnosis is confirmed. The patients will be followed up till discharge from hospital or 30 days after start of antifungal therapy or death (whichever is earlier).

6.3 Data collection - The form (Annexure II) will be filled up within 5 days of diagnosis of candidemia. The investigator would make sure that the patient is not identified (No mention of patient's name, address, hospital registration no. or any laboratory no. on the survey forms). The data collection will be performed both on line and on hard copy. The following variable will be noted:

1. Demographic data
2. Evaluation of the severity of the patient (severity will be assessed on the basis of scoring system available in the hospital (e.g, APACHE, SOFA).
3. Underlying disease
4. Risk factors
5. History of previous antifungal therapy (prophylaxis/empiric/ definitive treatment)
6. Description of candidemia episode
7. Laboratory results
8. Diagnosis of candidemia. 6.4 Laboratory or mycological tests - No laboratory or microbiological test is mandatory for the patient as a part of study. Study protocol will not intervene anywhere in laboratory investigation of the patient. Data of the laboratory tests performed as part of routine will be collected on study cases forms 6.5 Patient management: The study will not intervene anywhere in patient management. The clinician in charge will manage the patient. The data of management practiced will be incorporated retrospectively in management form (Annexure III) within 7 days of patient's discharge from hospital or 30 days after start antifungal therapy or patient's death (whichever is earlier) 6.6 Identification of Candida isolates and antifungal susceptibility testing: Candida isolates may be identified and antifungal susceptibility testing may be performed at the study centers as part of the center's routine procedure. However, all Candida isolates (isolated from blood) will be submitted to the reference laboratory at Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh after filling the form IV. PGIMER, Chandigarh will confirm the identity of all Candida isolates and perform antifungal susceptibility testing according to CLSI M27-A3 protocol (broth microdilution method) 6.7. Statistical analysis: Descriptive statistical methods will be employed to analyze the data.

7. Security and Confidentiality Once the patient is deemed eligible to participate and consent has been obtained (if any), a unique study number will be assigned. Subject initials and institution identification will be entered into a log book that will remain sole property of each site. The logbook will be kept secured at each site according to site's policies and procedures. The logbook will assist the investigator at the particular Institute to track and upload data in the system. Each site will be able to view its own patients entered and summary data on the aggregate patients of all centers, but no data from other sites.

8. Publication : In the event of publication, the Investigators' names that will be cited will be those who have attributed the largest number of cases of the study. The coordinator and the advisor will also be cited. The order of the authorship would depend upon the number of cases per investigator per center, in the decreasing order. The exact number of authors remains to be decided upon, but the maximum number may be restricted to 11. The 'SIHAM' candidemia network will be mentioned at the end of authors. All other investigators will be acknowledged as participants of the network in the appendix. The sponsor of the network will be acknowledged in each publication. None of the sites is permitted to make any publication on its sites data, based solely on the parameters included in this study for the cases included in the present study, during this study period. If there is any breach of this understanding, the data from that centre will not be included in the final data analysis.

9. Ethical Issue: The project should be cleared by the participating centers at their respective local Ethics Committee before commencing the project. The Ethics approval Certificate should be submitted to the coordinator before commencing the project.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in ICUs for > 48 hour
* All age group patients will be included (both adult & children)
* Diagnosed as proven candidemia with isolation of Candida species ≥1 occasion from blood during ICU stay.
* Blood culture positive for Candida spp. , if sample has been drawn within 48 hrs after discharge from the ICU.

Exclusion Criteria:

* Patient already diagnosed for candidemia before admission in ICUs or in ICU for ≤48h .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with candidemia diagnosed in ICUs > 48 h after admission during the study period will be included in each site
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Death or discharge | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Arunaloke Chakrabarti, MD, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- Arunaloke Chakrabarti, Chandigarh, Uttarakhand, India